CLINICAL TRIAL: NCT04613388
Title: Multicenter Registry Study on Proton Radiotherapy for Mediastinal Lymphomas
Brief Title: Registry Study of Proton Radiotherapy in Lymphoma
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Other Study IDs: RadOnk 130718
Record Dates: First submitted 2020-10-15; First posted 2020-11-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Mediastinal Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assesment of Effectiveness and side effects — Case Report forms, Quality of life questionaire

SUMMARY:
The aim is to record and document a mediastinal PT and the corresponding follow-up data (effectiveness and side effects). General recommendations for planning and feasibility are made within the framework of this study.

DETAILED DESCRIPTION:
Improvements in multimodal therapy have resulted in high curation rates in lymphoma patients. In addition, these cancer entities (Hodgkin lymphoma and non-Hodgkin lymphoma) often affect very young patients. Due to the high healing rates, the long-term effects of therapy are increasingly coming into focus: more than 40% of patients suffer from chronic, therapy-associated secondary diseases 30 years after successful therapy [1]. For this reason, an important focus of current research is the reduction of therapy-associated toxicity. A certain trend of dose reduction and reduction of the radiation fields (involved-field, involved-node, involved-site radiation) can already be seen in the research results of the last decades. Another interesting approach to protecting adjacent organs is the use of modern radiation techniques such as particle therapy with protons (PT).

In the case of radiation in the mediastinal area in particular, the use of PT can greatly reduce the dose in the area of the heart muscle, the lungs or the mammary gland tissue compared to conventional radiation with photons. It is hoped that this will result in a decrease, especially in chronic side effects, in the area of these organs. Since this is a group of young patients with intensive pre-treatment with chemotherapeutic agents, a reduction in long-term toxicities is of particular importance. In particular, cardiac and pulmonary long-term side effects as well as a reduction in the secondary malignancy rate play a major role in this collective.

The aim of this prospective registry study on proton radiotherapy for mediastinal lymphomas is to record the frequency, feasibility and side effects after PT in this group of patients. These data should then serve as the basis for concrete therapy recommendations and assessment of side effects. Close cooperation with the study groups should also enable a comparative analysis of comparable patients who were not treated with protons at a later point in time.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed lymphoma according to WHO

* Patient consent
* Patient age ≥18 years.
* Presence of the need for mediastinal radiotherapy and the presumed benefit of mediastinal radiotherapy using protons in comparison to photon radiation (e.g. improved heart, lungs, and breast protection compared to photon radiation).
* Ability of the patient to give consent

Exclusion Criteria:

Age <18 years

* Non-consent of the patient to the disclosure of his data
* Cancellation of the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mediastinal lymphoma are recorded who require consolidating mediastinal radiotherapy as part of their primary therapy. Since there is no intervention in the registry study, patients who are being treated in a therapy study (e.g. in the context of the ongoing Hodgkin studies) can also be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Acquisition and documentation of a mediastinal PT and the corresponding follow-up data | From date of written informed consent until the date of death from any cause, assessed up to 100 month
  Effectiveness and side effects of proton radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Laila König, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No